CLINICAL TRIAL: NCT02026700
Title: Bariederm Cream in Chronic Contact Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, rliranoHMO, DR, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bariederm-HMO-CTIL
Record Dates: First submitted 2013-12-22; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bariederm, barrier cream (Experimental): one arm study: use of bariederm cream on hands twice daily for 21 days
  Interventions: Device: bariederm cream

INTERVENTIONS:
Device: bariederm cream — patients are asked to apply twice a day a barrier cream on their hands for 3 weeks only
  Other Names: use of bariederm cream on hands twice daily for 21 days

SUMMARY:
We intend to evaluate the efficiency and tolerability of a barrier cream (bariederm) in protecting hands of individuals with hand dermatitis, either due to allergy or irritation. We believe that the use of the cream would benefit with the skin.

DETAILED DESCRIPTION:
The aim of the study is the evaluation of the effectiveness, tolerance and cosmetic acceptability of Bariéderm cream among patients presenting with chronic allergic or irritant contact dermatitis of the hands. We shall enrol adults presenting with CONTACT DERMATITIS EXCLUDING FLARE-UPS of the hands: whether allergic or irritant, able to understand the protocol and agrees to sign the information and informed consent form. Bariéderm cream will be applied minimum twice daily over 21 days. Response will be evaluated by self and physician filled questionnaires. effectiveness, tolerance and cosmetic acceptability will be evaluated by a scale of 1-10, 1 meaning "not at all" and 10 meaning "very much". Statistics will be performed by SPSS software with suitable statistical tests. In case of an adverse event caused by the product, patch-test with ingredients of Bariéderm cream will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients with dermatitis of the hands

Exclusion Criteria:

* pregnant ladies,
* known allergy to ingredients -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
self evaluation of effectiveness and tolerance in a 1-10 scale | 21 days
  effectiveness tolerance and acceptability in adults with hand dermatitis, evaluated by a self reported and a physician reported questionaires, using a 1-10 scale for evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Liran Horev Yakir, MD, Principal Investigator — Dept of Dermatology, Hadassah Medical Center, Jerusalem 911201, Israel
Locations (1):
- : Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel